CLINICAL TRIAL: NCT04713891
Title: A Phase I, Multi-Center, Open-Label Study to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Anti-tumor Activity of KF-0210 in Patients With Advanced Solid Tumors
Brief Title: A Study of KF-0210 in Advanced Solid Tumors Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keythera Pharmaceuticals (Australia) Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Keythera (Suzhou) Pharmaceuticals Co. Ltd (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KFCS001
Record Dates: First submitted 2020-11-25; First posted 2021-01-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumor; Colorectal Cancer; Lung Cancer; Squamous Cell Carcinoma of the Esophagus; Gastric Cancer; Bladder Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Esophageal Squamous Cell Carcinoma; Stomach Neoplasms; Urinary Bladder Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Phase 1a: Cohort 1 (Experimental): KF-0210 tablet will be administered at 120 mg as a single agent orally once daily (QD) continuously in cycles (1 cycle=21 days) until the disease progression, intolerance, or informed consent withdrawal.
  Interventions: Drug: KF-0210 tablets, 120 mg
- Phase 1a: Cohort 2 (Experimental): KF-0210 tablet will be administered at 240 mg as a single agent orally once daily (QD) continuously in cycles (1 cycle=21 days) until the disease progression, intolerance, or informed consent withdrawal.
  Interventions: Drug: KF-0210 tablets, 240 mg
- Phase 1a: Cohort 3 (Experimental): KF-0210 tablet will be administered at 450 mg as a single agent orally once daily (QD) continuously in cycles (1 cycle=21 days) until the disease progression, intolerance, or informed consent withdrawal.
  Interventions: Drug: KF-0210 tablets, 450 mg
- Phase 1a: Cohort 4 (Experimental): KF-0210 tablet will be administered at 600 mg as a single agent orally once daily (QD) continuously in cycles (1 cycle=21 days) until the disease progression, intolerance, or informed consent withdrawal.
  Interventions: Drug: KF-0210 tablets, 600 mg
- Phase Ib, Cohort 1 (Experimental): KF-0210 (dose RP2D-2, orally once daily)+ Atezolizumab (1200 mg every 3 weeks) continuously until disease progression/recurrence or death from any cause, or serious adverse events (SAE) observed (whichever occurs earlier) for up to 2 years.
  Interventions: Drug: KF-0210 (dosage RP2D-2) + Atezolizumab
- Phase Ib, Cohort 2 (Experimental): KF-0210 (dose RP2D-1, orally once daily)+ Atezolizumab (1200 mg every 3 weeks) continuously until disease progression/recurrence or death from any cause, or serious adverse events (SAE) observed (whichever occurs earlier) for up to 2 years.
  Interventions: Drug: KF-0210 (dosage RP2D-1) + Atezolizumab
- Phase Ib, Cohort 3 (Experimental): KF-0210 (dose RP2D, orally once daily)+ Atezolizumab (1200 mg every 3 weeks) continuously until disease progression/recurrence or death from any cause, or serious adverse events (SAE) observed (whichever occurs earlier) for up to 2 years.
  Interventions: Drug: KF-0210 (dosage RP2D) + Atezolizumab

INTERVENTIONS:
Drug: KF-0210 tablets, 120 mg — KF-0210 tablet will be orally administered as a single agent at 120 mg once daily (QD) continuously, until the disease progression, intolerance, or informed consent withdrawal.
  Other Names: KF-0210-0
  Arms: Phase 1a: Cohort 1
Drug: KF-0210 tablets, 240 mg — KF-0210 tablet will be orally administered as a single agent at 240 mg once daily (QD) continuously, until the disease progression, intolerance, or informed consent withdrawal.
  Other Names: KF-0210-0
  Arms: Phase 1a: Cohort 2
Drug: KF-0210 tablets, 450 mg — KF-0210 tablet will be orally administered as a single agent at 450 mg once daily (QD) continuously, until the disease progression, intolerance, or informed consent withdrawal.
  Other Names: KF-0210-0
  Arms: Phase 1a: Cohort 3
Drug: KF-0210 tablets, 600 mg — KF-0210 tablet will be orally administered as a single agent at 600 mg once daily (QD) continuously, until the disease progression, intolerance, or informed consent withdrawal.
  Other Names: KF-0210-0
  Arms: Phase 1a: Cohort 4
Drug: KF-0210 (dosage RP2D-2) + Atezolizumab — KF-0210 tablet will be orally administered at dosage RP2D-2 once daily (QD) in combination with Atezolizumab that will be administered at 1200 mg every 3 weeks via intravenously infusion.
  Other Names: KF-0210-0; Tecentriq
  Arms: Phase Ib, Cohort 1
Drug: KF-0210 (dosage RP2D-1) + Atezolizumab — KF-0210 tablet will be orally administered at dosage RP2D-1 once daily (QD) in combination with Atezolizumab that will be administered at 1200 mg every 3 weeks via intravenously infusion.
  Other Names: KF-0210-0; Tecentriq
  Arms: Phase Ib, Cohort 2
Drug: KF-0210 (dosage RP2D) + Atezolizumab — KF-0210 tablet will be orally administered at dosage RP2D once daily (QD) in combination with Atezolizumab that will be administered at 1200 mg every 3 weeks via intravenously infusion.
  Other Names: KF-0210-0; Tecentriq
  Arms: Phase Ib, Cohort 3

SUMMARY:
The purpose of this Phase I, Multi-Center, Open-Label Study is to evaluate the safety, tolerability, Pharmacokinetics, Pharmacodynamics and anti-tumor activity of KF-0210 in participants with advanced solid tumors. The study will be conducted in two parts: phase Ia, and phase Ib.

DETAILED DESCRIPTION:
Phase 1a:

The primary objective of the phase 1a part of the study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamic and anti-tumor activity of oral KF-0210 as a single agent in participants with advanced solid tumors, to identify the dose-limiting toxicity and establish the maximum tolerated dose, or maximum administered dose and/or the recommended Phase II dose of KF-0210 in participants with advanced solid tumors.

Phase 1b:

The primary objective of the phase 1b part of the study is to assess the safety, pharmacokinetics, pharmacodynamic and anti-tumor activity of KF-0210 in combination with Atezolizumab in patients with colorectal cancer (CRC) (MSS), lung cancer (LC), squamous cell carcinoma of the esophagus (SCCE), gastric cancer (GC), and bladder cancer (BC).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male and female;
2. Patients are confirmed by available pathology records or current biopsy having advanced, nonresectable, or recurrent and progressing solid tumors since last anti-tumor therapy, and who are unavailable or intolerable for available standard therapy or there is no standard available therapy.

   * Phase Ia (Dose Escalation): Advanced solid tumors;
   * Phase Ib (Expansion Study): Patients must have any of the following tumor type and have not participated in Phase Ia trial of this study: CRC (MSS), LC, SCCE, GC, and BC. Among them, patients with LC, SCCE, or GC must have undergone PD-1/PD-L1 treatment for at least 12 weeks and failed.
3. Must have at least 1 measurable lesion, according RECIST V1.1 criteria (CT-scans or MRI no longer than 4 weeks before signing ICF);
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Life expectancy≥ 3 months;
6. Females must not be lactating or pregnant at screening or baseline (negative pregnant test).

Exclusion Criteria:

1. Patients with prior anti-tumor therapy within 4 weeks prior to first dosing of KF-0210, including chemotherapy, biotherapy, endocrine therapy and immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer);
2. Patients with prior definitive radiation therapy within 6 weeks prior to first dosing of KF-0210, and the irradiated lesions showed no signs of progression if it to be considered target lesions. Or patients with prior palliative radiotherapy within 2 weeks prior to first dosing of KF-0210. Or the radiotherapy-related side effects have unresolved before the study entry. Or use of radiopharmaceuticals (strontium, samarium) within 8 weeks prior to first dosing of KF-0210;
3. Patients who have another active malignancy which is likely to require treatment;
4. Patients who have known active central nervous system (CNS) metastases and/or carcinomatous meningitis;
5. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months prior to the first dose of KF-0210; or cardiac arrhythmia requiring medical treatment (including oral anticoagulation);
6. Patients with any active autoimmune disease or a documented history of autoimmune disease, poorly controlled asthma or history of syndrome that required systemic steroids or immunosuppressive medications, except for patients with vitiligo or resolved childhood asthma/atopy. Patients with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study;
7. Patients with inflammatory bowel disease or digestive tract diseases (e.g. peptic ulcer disease, including stomach and duodenal ulcer, gastritis and enteritis);
8. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of KF-0210;
9. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids except inhaled or intranasal corticosteroids (with minimal systemic absorption);
10. Current use of NSAIDs, COX-1/COX-2 inhibitors within 4 weeks;
11. Patients who have received surgical or interventional treatment (excluding tumor biopsy, puncture, etc.) within 28 days prior to first dosing of KF-0210;
12. Use of other investigational drugs within 28 days or at least 5 half-lives (whichever is shorter) prior to the first dosing of KF-0210;
13. Use of any live vaccines (e.g., intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines) within 28 days prior to the first dosing of KF-0210;
14. Any unresolved toxicities from prior therapy, greater than Common Terminology Criteria for Adverse Events (CTCAE 5.0) grade 1 at the time of starting study treatment with exception of alopecia;
15. Any uncontrolled or severe illness, including but not limited to: ongoing or active infection requiring parenteral antibiotics;
16. Positive screening tests for any one of them: human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg); hepatitis B core antibody (HBcAb) (negative for HBsAg, but HBcAb positive, an HBV-DNA test will be performed and if positive will be excluded), hepatitis C antibody (anti-HCV positive, but negative HCV RNA test is allowed to be included).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Percentage of patient with adverse events / serious adverse events (AEs/SAEs) [Safety and Tolerability] | From consent through 28 days (±7 days) after the last dose or before starting other anti-tumor treatment (whichever occurs earlier)(up to approximately 1 year))
  Adverse events will be assessed according to CTCAE V5.0, and be coded according to the MedDRA Dictionary
Dose limiting toxicity (DLT) of KF-0210 [Tolerability] | From Cycle 1 Day 1 to Cycle 1 Day 21, each cycle is 21 days.
  Dose limiting toxicity (DLT) will be considered to be related to KF-0210 according to CTCAE V5.0 including hematology toxicities, non-hematological toxicities and any other toxicities.
Maximum tolerated dose (MTD) of KF-0210 alone [Tolerability] | Up to 21 days after first administration in cycle 1, each cycle is 21 days
  The Maximum tolerated dose (MTD) is defined as the highest dose at which ≤1、6 participants occurred dose limiting toxicity at each dose level.
Change of Body Weight from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 1 of each cycle (each cycle is 21 days), and at the end of treatment/withdrawal (up to approximately 1 year)
  Body Weight measured in kilogram (kg)
Change of Body Temperature from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  Axillary temperature measured in celsius
Change of Pulse rate from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  Pulse rate measured per minute
Change of Systolic pressure from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  Blood pressure measured in mmHg
Change of Diastolic pressure from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  Blood pressure measured in mmHg
Change of Heart rate from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  Heart rate in beats per minute (Bpm) through 12-lead ECG assessment
Change of R-R interval from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  R-R interval measured in millisecond through 12-lead ECG assessment
Change of P-R interval from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  P-R interval measured in millisecond through 12-lead ECG assessment
Change of QRS complex from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  QRS complex measured in millisecond through 12-lead ECG assessment
Chang of QT interval from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  QT interval measured in millisecond through 12-lead ECG assessment
Change of corrected QT (QTc) interval from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  corrected QT (QTc) interval measured in millisecond through 12-lead ECG assessment
Change of Fridericia's Correction QT (QTcF) interval from Baseline [Safety] | From screening to the end of treatment/withdrawal (up to approximately 1 year)
  Fridericia's Correction QT (QTcF) interval measured in millisecond through 12-lead ECG assessment.
Change of Eastern Cooperative Oncology Group-Performance Status (ECOG PS) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 1 of each cycle (each cycle is 21 days), and at the end of treatment/withdrawal (up to approximately 1 year)
  The performance status will be evaluated in accordance with the Eastern Cooperative Oncology Group (ECOG) criteria with the score range in 0 to 5. A score of 0 represents fully normal activity and a score of 5 represents death.
Change of Total Protein (TP) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Total Protein (TP) measured in g/dL
Change of Albumin (ALB) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Albumin(ALB) measured in g/dL
Change of Alanine aminotransferase (ALT) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Alanine aminotransferase (ALT) measured in IU/L
Change of Aspartate aminotransferase (AST) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Aspartate aminotransferase (AST) measured in IU/L
Change of Alkaline phosphatase (ALP/AKP) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Alkaline phosphatase (ALP/AKP) measured in IU/L
Change of Total bilirubin from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Total bilirubin measured in mg/dL
Change of Direct bilirubin from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Direct bilirubin measured in mg/dL
Change of Indirect bilirubin from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Indirect bilirubin measured in mg/dL
Change of Glutamyl transpeptidase from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Glutamyl transpeptidase measured in U/L
Change of Blood glucose from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Blood glucose measured in mg/dL
Change of Urea from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Urea measured in mg/dL
Change of Uric acid from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Uric acid measured in mg/dL
Change of Creatinine from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Creatinine measured in mg/dL
Change of Creatinine Kinase from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Creatinine Kinase measured in IU/L
Change of Total Cholesterol from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Total Cholesterol measured in mmol/L
Change of Triglycerides from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Triglycerides measured in mmol/L
Change of Potassium, Sodium, Chloride or Calcium from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Potassium, Sodium, Chloride or Calcium measured in mmol/dL
Change of Leukocyte Count from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Leukocyte Count measured in K/uL
Change of Neutrophil Count from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Neutrophil Count in K/uL
Change of Percentage of Neutrophil from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Percentage of Neutrophil will be measured
Change of Lymphocyte Count from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Lymphocyte Count measured in K/uL
Change of Percentage of Lymphocyte from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Percentage of Lymphocyte will be measured
Change of Monocytes Count from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Monocytes Count measured in K/uL
Change of Percentage of Monocytes from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Percentage of Monocytes will be measured
Change of Eosinophils Count from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Eosinophils Count measured in K/uL
Change of Percentage of Eosinophils from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Percentage of Eosinophils will be measured
Change of Basophil Count from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Basophil Count measured in K/uL
Change of Percentage of Basophil from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Percentage of Basophil will be measured
Change of Erythrocyte Count from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Erythrocyte Count measured in K/uL
Change of Hemoglobin from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Hemoglobin measured in mg/dL
Change of Hematocrit Platelets from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Hematocrit Platelets measured in K/uL
Change of Coagulation test-Activated partial thromboplastin time (APTT) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Activated partial thromboplastin time (APTT) measured in seconds
Change of Coagulation test-Prothrombin time (PT) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Prothrombin time (PT) measured in seconds
Change of Coagulation test-Fibrinogen(FIB) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Fibrinogen(FIB) measured in mmol/L
Change of Coagulation test-Thrombin time (TT) from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Thrombin time (TT) measured in seconds
Change of Urine pH from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  pH value will be measured
Change of Specific gravity of urine from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Specific gravity value will be measured
Change in Occult blood result from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  The result will be recorded as either positive or negative
Change in Urine Bilirubin result from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Urine bilirubin will be measure in µmol/L
Change in Urine protein from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Urine protein will be measured in mg/dL
Change in Urine Glucose from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Urine Glucose will be measured in mg/dL
Change in Ketones from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Ketones will be measured in mg/dL
Change in Urobilinogen from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Urobilinogen will be measured in EU/dL
Change in Urinary leukocyte from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Urinary leukocyte will be counted in K/uL
Change in Urine erythrocytes from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Urine erythrocytes will be counted in K/uL
Change in Urine Nitrites from Baseline [Safety] | On date of screening (within 7 days before the first dose), Day 8, Day15, Day 21 of cycle 1 (each cycle is 21 days), Day 1 of each cycle from the cycle 2, and at the end of treatment/withdrawal (up to approximately 1 year)
  Urobilinogen will be measured in mg/dL
Clinically significant abnormality in physical examinations | On date of screening (within 7 days before the first dose), Day 1 of each cycle (each cycle is 21 days), and at the end of treatment/withdrawal (up to approximately 1 year)
  Physical examination includes skin, head, eyes, ears, nose and throat, lymph nodes, heart, chest, abdomen and extremities, and nervous system (speech, cranial nerves, motor ability, tendon reflexes, sensations, free movement)

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Phase I a: specific time points from Cycle 1 Day 1 to Cycle 1 Day 8; Phase 1b: specific time points from Cycle 1 Day 1 to Cycle 4 Day 5, each cycle is 21 days.
  For KF-0210 alone in phase Ia, and for KF-0210 and Atezolizumab in Phase Ib. Calculated by non-compartmental analysis (NCA) for WinNonlin V8.2 (or above).
Time of maximum plasma concentration (Tmax) | Phase I a: specific time points from Cycle 1 Day 1 to Cycle 1 Day 8; Phase 1b: specific time points from Cycle 1 Day 1 to Cycle 4 Day 15. Each cycle is 21 days.
  For KF-0210 alone in phase Ia, and for KF-0210 and Atezolizumab in Phase Ib. Calculated by non-compartmental analysis (NCA) for WinNonlin V8.2 (or above).
Area under the plasma concentration-time curve from time-zero extrapolated to infinite time (AUC0-inf) | Phase I a: specific time points from Cycle 1 Day 1 to Cycle 1 Day 8; Phase 1b: specific time points from Cycle 1 Day 1 to Cycle 4 Day 15. Each cycle is 21 days.
  For KF-0210 alone in phase Ia, and for KF-0210 and Atezolizumab in Phase Ib. Calculated by non-compartmental analysis (NCA) for WinNonlin V8.2 (or above).
Area under the plasma concentration-time curve from time-zero to the time of the last measurable concentration (AUC0-t) of KF-0210 | Phase I a: specific time points from Cycle 1 Day 1 to Cycle 1 Day 8; Phase 1b: specific time points from Cycle 1 Day 1 to Cycle 4 Day 15. Each cycle is 21 days.
  For KF-0210 alone in phase Ia, and for KF-0210 and Atezolizumab in Phase Ib. Calculated by non-compartmental analysis (NCA) for WinNonlin V8.2 (or above).
Terminal half-life (T1/2) of KF-0210 | Phase I a: specific time points from Cycle 1 Day 1 to Cycle 1 Day 8; Phase 1b: specific time points from Cycle 1 Day 1 to Cycle 4 Day 15. Each cycle is 21 days.
  For KF-0210 alone in phase Ia, and for KF-0210 and Atezolizumab in Phase Ib. Calculated by non-compartmental analysis (NCA) for WinNonlin V8.2 (or above).
Accumulation ratio (Rac) | Phase I a: specific time points from Cycle 1 Day 1 to Cycle 1 Day 8; Phase 1b: specific time points from Cycle 1 Day 1 to Cycle 4 Day 15. Each cycle is 21 days.
  For KF-0210 alone in phase Ia, and for KF-0210 and Atezolizumab in Phase Ib. Calculated by non-compartmental analysis (NCA) for WinNonlin V8.2 (or above).
Cmin to Cmax fluctuation between dose time and Tau (DF) | Phase I a: specific time points from Cycle 1 Day 1 to Cycle 1 Day 8; Phase 1b: specific time points from Cycle 1 Day 1 to Cycle 4 Day 15. Each cycle is 21 days.
  For KF-0210 alone in phase Ia, and for KF-0210 and Atezolizumab in Phase Ib. Calculated by non-compartmental analysis (NCA) for WinNonlin V8.2 (or above).
Blood cytokines/chemokines levels | Up to 21 days after first administration in cycle 1, each cycle is 21 days.
  Biomarker for pharmacodynamic assessment including interferon (IFN-γ), tumor necrosis factor (TNF-α), CXCL10 and CCL5.
Urine prostaglandin metabolites level | Up to 21 days after first administration in cycle 1, each cycle is 21 days.
  To explore the prostaglandin metabolites in urine
Tumor T cell infiltration | Up to 21 days after first administration in cycle 1, each cycle is 21 days.
  Tumor biopsies will be analyzed by immunohistochemistry (IHC) for CD3+ T cells, CD8+ T cells and PD-L1 expression.
Change in tumor size from baseline | From screening through the last dose of treatment, each cycle is 21 days.
  Tumor assessment with CT scan or MRI. The anti-tumor activity will be evaluated according to the RECIST V1.1.
Objective response rate (ORR) | From screening through the last dose of treatment, each cycle is 21 days.
  Tumor assessment with CT scan or MRI. The tumor lesions will be evaluated according to the RECIST V1.1 standard, and categorized into complete response(CR), partial response (PR), stable disease (SD) , and progressive disease (PD).
Duration of response (DOR) (days) | From screening through the last dose of treatment, each cycle is 21 days.
  Tumor assessment with CT scan or MRI. The tumor lesions will be evaluated according to the RECIST V1.1 standard, and categorized into complete response(CR), partial response (PR), stable disease (SD) , and progressive disease (PD).
Disease control rate (DCR) | From screening through the last dose of treatment, each cycle is 21 days.
  Tumor assessment with CT scan or MRI. The tumor lesions will be evaluated according to the RECIST V1.1 standard, and categorized into complete response(CR), partial response (PR), stable disease (SD) , and progressive disease (PD).
Progression free survival (PFS) | From screening through the last dose of treatment, each cycle is 21 days.
  Tumor assessment with CT scan or MRI. The tumor lesions will be evaluated according to the RECIST V1.1 standard, and categorized into complete response(CR), partial response (PR), stable disease (SD) , and progressive disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Cosman, MD, Principal Investigator — Scientia Clinical Research Ltd
Locations (1):
- Scientia Clinical Research Limited, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No